CLINICAL TRIAL: NCT05590780
Title: Analysis of the Impact of Cell-free DNA (cfDNA) During Periodontitis and Cardiovascular Disease
Brief Title: Analysis of Cell-free DNA (cfDNA) During Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Other Study IDs: 121/20/22/PO
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Periodontal Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Evaluation of plasma cfDNA levels
  Interventions: Other: Clinical Attachment level
- Periodontitis: Evaluation of plasma cfDNA levels
  Interventions: Other: Clinical Attachment level
- Cardiovascular disease: Evaluation of plasma cfDNA levels
  Interventions: Other: Clinical Attachment level
- Periodontitis + cardiovascular disease: Evaluation of plasma cfDNA levels
  Interventions: Other: Clinical Attachment level

INTERVENTIONS:
Other: Clinical Attachment level — 1-year
  Other Names: Evaluation of changes (in millimeters) of Clinical attachment level loss

SUMMARY:
The purpose of this study was to examine the association between circulating cfDNA concentration and CVD risk in patients with periodontitis, CVD, and periodontitis plus CVD. In addition, the secondary objective was to identify, among other confounders, the impact of periodontitis and cardiovascular disease as potential significant predictors of circulating cfDNA levels in the enrolled population.

DETAILED DESCRIPTION:
Recent emerging evidence has shown that circulating cell-free (cf) DNA are involved in in several epigenetic processes linked with periodontitis, coronary stenosis and systemic inflammation. The present study was aimed at assessing the impact of periodontitis on circulating cfDNA levels and evaluating possible confounders that influenced this association. Healthy controls (n=30) and subjects with CVD (n=31), periodontitis (n=31) and periodontitis+CVD (n=30) were enrolled. All subjects underwent regular periodontal examination and blood sampling. The analysis of the plasma cfDNA concentrations was performed using a dsDNA Assay Kit.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 15 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy controls (n=30) and subjects with CVD (n=31), periodontitis (n=31) and periodontitis+CVD (n=30) were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level loss | baseline changes
  Evaluation of changes (in millimeters) of Clinical attachment level loss
circulating cell-free DNA | baseline changes
  Evaluation of changes (in millimeters) of plasma circulating cell-free DNA

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- University of Catania, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Undecided
all collected IPD, all IPD that underlie results in a publication